CLINICAL TRIAL: NCT02350439
Title: Differential Effect of High (200μg/kg/Min) Adenosine Dose on Fractional Flow Reserve in Patients Presenting Variation of FFR ≥0.05 During the Usual Dose of Adenosine Infusion (140μg/kg/Min).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor, University of Patras
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PATRASCARDIOLOGY 19
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Fractional floe reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adenosine intravenous infusion at 200μg/Kg/min (Experimental): Fractional flow reserve assessment under Adenosine intravenous infusion at 200μg/Kg/min
  Interventions: Drug: Adenosine infusion at 200μg/Kg/min

INTERVENTIONS:
Drug: Adenosine infusion at 200μg/Kg/min — Assessment of fractional flow reserve (FFR) under high adenosine intravenous infusion dose (200mg/kg/min)

SUMMARY:
Fractional flow reserve (FFR) is an established invasive method for assessing the physiological significance of coronary artery stenosis. However, in recent studies it has been observed and reported some degree of variation in the fraction of the coronary artery to the aortic pressure (Pd / Pa) during the infusion of standard adenosine dose (140mg/kg/min). The observed variation may be attributed to a failure to achieve maximal hyperemia with the normal dose. The administration of adenosine at a higher dose (200μg/kg /min) may influence coronary flow reserve (FFR) eliminating Pd / Pa variation during adenosine infusion.

This is a prospective study which will be conducted in patients after coronary angiography with at least one angiographic lesion ≥50% in coronary vessels.

Patients after written consent will undergo assessment of lesion severity with FFR under a three-minute infusion of adenosine 140mg/kg/min. In patients during steady state hyperaemia (determined by visual assessment) exhibiting variation in Pd / Pa ratio ≥ 0.05 (e.g. difference of max Pd/Pa minus min Pd/Pa) the examination will be repeated after 5 min with three-minute infusion under high dose adenosine (200mg/kg/min). The minimum ratio Pd/Pa per 3 beats will be offline analyzed. The FFR during steady hyperemia state is defined as the average of the minimum ratio Pd / Pa per three beats.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. Patients with at least 1 ≥50% stenosis in a coronary vessel, subjected to FFR assessment, who exhibit variation in Pd / Pa ratio ≥ 0.05 (e.g. difference of max Pd/Pa minus min Pd/Pa) during steady state hyperaemia (determined by visual assessment).
3. Written informed consent

Exclusion Criteria:

1. Left main disease (angiographically> 50%)
2. Cardiogenic shock / hemodynamic instability
3. Previous CABG
4. Increased risk of bradycardia on investigator clinical judgment
5. Severe chronic obstructive pulmonary disease
6. Coronary vessels with tortuosity or extremely calcified
7. Severe left ventricular hypertrophy or severe valvular disease
8. STEMI or non-STEMI within the past five days
9. Previous myocardial infarction in the distribution of the target vessel for the FFR
10. Acute decompensated heart failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Difference between the maximum and minimum value of Pd / Pa ratio during steady state hyperaemia between the 2 groups. | 10 minutes
Coefficient of variation of Pd / Pa ratio during steady state hyperemia between the 2 groups | 10 minutes

SECONDARY OUTCOMES:
FFR value as determined by the software, between the 2 groups. | 10 minutes
FFR during steady state hyperemia. | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Patras University Hospital, Pátrai, Greece

REFERENCES:
- [Derived] Alexopoulos D, Xanthopoulou I, Tsigkas G, Koutsogiannis N, Salata P, Armylagos S, Moulias A, Davlouros P. Effect of High (200 mug/kg per Minute) Adenosine Dose Infusion on Fractional Flow Reserve Variability. J Am Heart Assoc. 2016 Nov 10;5(11):e004323. doi: 10.1161/JAHA.116.004323. PMID 27930357